CLINICAL TRIAL: NCT04810598
Title: Evaluation of the Pharmacokinetics and Safety of Venetoclax in Subjects With Impaired Renal Function
Brief Title: Study to Assess Adverse Events and the Movement of Oral Venetoclax Tablet Through the Body of Female Participants Aged 18-75 Years With Impaired Renal Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Collaborators: Roche-Genentech (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: M19-065
Record Dates: First submitted 2021-03-19; First posted 2021-03-23 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2022-09

CONDITIONS: Renal Impairment; Renal Disease
Keywords: Renal Impairment; Renal Disease; End stage renal disease (ESRD); Venetoclax; Venclexta
MeSH Terms: conditions — Renal Insufficiency; Kidney Diseases; Kidney Failure, Chronic | interventions — venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group 1: Participants With Normal Renal Function (Experimental): Participants with normal renal function will receive single dose of venetoclax on Day 1.
  Interventions: Drug: Venetoclax
- Group 2: Participants With End Stage Renal Disease (Experimental): Participants with end stage renal disease (ESRD) will receive single dose of venetoclax on Period 1 Day 1 and Period 2 Day 1 (Each period is 3 days separated by 7-day washout period).
  Interventions: Drug: Venetoclax

INTERVENTIONS:
Drug: Venetoclax — Oral Tablet
  Other Names: Venclexta; ABT-199; GDC-0199

SUMMARY:
Renal insufficiency is common in participants with blood cancers. The main objective of this study is to evaluate adverse events and movement of oral venetoclax tablets through the body of female participants with severe normal renal function and those with end stage renal disease (ESRD) requiring hemodialysis.

Venetoclax is an investigational drug being developed for the treatment of various hematologic malignancies. Study doctors put the participants in 1 of 2 groups, called treatment arms. Each group receives a different treatment. Approximately 12 female participants between 18 and 75 years, with Body Mass Index (BMI) between 18 to 42 kg/m2 will be enrolled in approximately 4 sites across the world.

Participants with normal renal function will receive single dose of oral venetoclax tablet. Participants with ESRD will receive oral venetoclax tablets just prior to hemodialysis (Period 1 Day 1) and between dialysis days (Period 2 Day 1), doses in the two periods will be separated by at least 7 days.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, blood and urine tests, checking for side effects.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) between 18.0 and 42.0 kg/m2.
* Postmenopausal or permanently surgically sterile (bilateral oophorectomy, bilateral salpingectomy, or hysterectomy).
* Women of childbearing potential, practicing at least 2 protocol specified methods of birth control that are effective from at least 30 days before starting study drug through at least 30 days after the last dose of any study drug.
* Group 1 only: Must be in general good health based upon the results of a medical history, physical examination, and 12-lead electrocardiogram (ECG) with normal Glomerular Filtration Rate (GFR) at Screening.
* Group 2 only: Stable condition and acceptable for study participation based upon the results of a medical history, physical examination, laboratory profile, and ECG. Participant with end stage renal disease (ESRD) requiring dialysis on hemodialysis must have been receiving hemodialysis for at least 1 month.

Exclusion Criteria:

- Participants on a strict vegetarian or vegan diet.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-07-08 (Actual); Primary Completion 2022-08-16 (Actual); Study Completion 2022-08-16 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With Adverse Events (AEs) | Up to approximately 38 days
  An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment. The investigator assesses the relationship of each event to the use of study. A serious adverse event (SAE) is an event that results in death, is life-threatening, requires or prolongs hospitalization, results in a congenital anomaly, persistent or significant disability/incapacity or is an important medical event that, based on medical judgment, may jeopardize the participant and may require medical or surgical intervention to prevent any of the outcomes listed above.
Maximum Plasma Concentration (Cmax) of Venetoclax (Groups 1,2) | Up to Day 6
  Maximum Plasma Concentration (Cmax) of Venetoclax.
Time to Cmax (Tmax) of Venetoclax (Groups 1,2) | Up to Day 6
  Time to Cmax (Tmax) of Venetoclax.
Area Under the Plasma Concentration-time Curve over time from time 0 to 48 hours (AUC0-48) of Venetoclax (Groups 1,2) | Up to Day 6
  Area Under the Plasma Concentration-time Curve over time from time 0 to 48 hours (AUC0-48).
Pre-dose Unbound Fraction (fu) of Venetoclax in Plasma (Groups 1,2) | Day 1
  Unbound Fraction (fu) of Venetoclax in Plasma.
Dialysis Clearance (CLdialysis) (Group 2) | Day 1
  Dialysis Clearance (CLdialysis) is calculated in participants undergoing hemodialysis in Period 1.
Unbound Fraction Pre-dialysis (fu,predialysis) of Venetoclax in Plasma (Group 2) | Day 1
  Unbound fraction pre-dialysis (fu,predialysis) of venetoclax in plasma is calculated in participants undergoing hemodialysis in Period 1.
Unbound Fraction Post-dialysis (fu,postdialysis) of Venetoclax in Plasma (Group 2) | Day 1
  Unbound fraction post-dialysis (fu,postdialysis) of venetoclax in plasma is calculated in participants undergoing hemodialysis in Period 1.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (2):
- United States (2):
  - Orlando Clinical Research Ctr /ID# 224922, Orlando, Florida
  - Acpru /Id# 243398, Grayslake, Illinois

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: This clinical study may be evaluating a usage that is not currently FDA approved. Please see US Prescribing Information for approved uses. — https://www.rxabbvie.com/